CLINICAL TRIAL: NCT06727812
Title: A Phase I Clinical Study of the Safety, Tolerability, Pharmacokinetics, and Initial Efficacy of HRS-6208 Monotherapy in Patients With Advanced Solid Tumors
Brief Title: Multicenter Phase I Study of HRS-6208 in Patients With Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-6208-101
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental)
  Interventions: Drug: HRS-6208

INTERVENTIONS:
Drug: HRS-6208 — HRS-6208.

SUMMARY:
This is an open, multicenter Phase I study to evaluate the safety and tolerability of HRS-6208 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unresectable locally advanced or metastatic solid tumors confirmed by histology or cytology who have relapsed or progressed after standard treatment, or have no standard treatment options, or do not apply standard treatment at this stage;
2. Age 18~75 years old;
3. At least one measurable lesion per RECIST v1.1 criteria;
4. ECOG PS score: 0-1.

Exclusion Criteria:

1. History of other malignancies within the past 5 years, excluding cured basal cell carcinoma of the skin and carcinoma in situ of the cervix;
2. The adverse reactions of previous anti-tumor therapy have not recovered to NCI-CTCAE v5.0 grade evaluation ≤ 1;
3. He has severe cardiovascular and cerebrovascular diseases;
4. Severe infection within 4 weeks prior to the first dose.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | From Day 1 to 30 days after the last dose.
Maximum tolerated dose (MTD) | From Day 1 to 21 days after the first dose.
Dose limiting toxicity (DLT) | From Day 1 to 21 days after the first dose.
Recommended phase 2 dose (RP2D) | From Day 1 to 30 days after the last dose.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From time of first dose of HRS-6208 until the date of objective disease progression or death (up to 24 months).
Duration of Response (DoR) | From time of first dose of HRS-6208 until the date of objective disease progression or death (up to 24 months).
Disease Control Rate (DCR) | From time of first dose of HRS-6208 until the date of objective disease progression or death (up to 24 months).
Progression free Survival (PFS) | From time of first dose of HRS-6208 until the date of objective disease progression or death (up to 24 months).
Overall Survival (OS) | From time of first dose of HRS-6208 until the date of objective disease progression or death (up to 24 months).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - West China Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided